CLINICAL TRIAL: NCT05510765
Title: ACTiN and Health Metrics: Improving Transportation Assets as a Critical Social Determinant of Health and the Effects on Wellness and Chronic Disease Metrics.
Brief Title: Improving Transportation Assets and the Effects on Wellness Metrics
Acronym: ACTiN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: John M. Salmon IV, MD (Other)
Responsible Party: Sponsor-Investigator, John M. Salmon IV, MD, Medical Director, Lighthouse Community Health Center, Unified Potential, Inc.
Organization: Unified Potential, Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4212.081022
Record Dates: First submitted 2022-08-10; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Social Determinants of Health
MeSH Terms: interventions — Transportation

STUDY DESIGN:
Intervention Model Description: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Low resource, high risk individuals with limited transportation options as a social determinant of health.
  Interventions: Behavioral: Transportation service

INTERVENTIONS:
Behavioral: Transportation service — Improved transportation assets applied to all aspects of subjects life

SUMMARY:
1. Implementation of an Advanced Connected Transportation Network (ACTiN), a novel, collaborative multinetwork transportation model for small cities and rural areas.
2. Evaluation of effectiveness in improving transportation assets for clients of a community-based nonprofit specializing in addressing social determinants of health (Lighthouse Community Health Services in Lynchburg, VA).
3. Simultaneous evaluation of wellness metrics based on the standards of the CMS Annual Wellness Visit and metrics associated with common chronic diseases.

DETAILED DESCRIPTION:
1. Implementation of a community transportation solution The project will be managed by Unified Potential, Inc., a 501c3 tax-exempt organization for transportation.

   * The solution requires implementation of four separate transportation "networks"
   * Public / Contracted / For-Hire Transportation
   * Workforce Transportation Network
   * Community Rideshare Network
   * Volunteer Transportation Network
2. Assessment of Personal Transportation Assets

   * Subjects asked to complete a survey upon intake, at six months, and at one year
   * Digital survey:
   * Can be completed by individual using provided smartphone app or at onsite desktop kiosk
   * Can be facilitated by a caregiver or other provider not involved in data analysis
3. Assessment of health and wellness metrics and chronic disease metrics if applicable

   * Dataset based on metrics assessed in the Center for Medicare and Medicaid Services (CMS) Annual Wellness Visit
   * All metrics quantified via either binary (yes/no) or through use of a validated scale (see below)
   * Data collected electronically at onsite or in-home provider visits at intake, six months, and one year

ELIGIBILITY:
Inclusion Criteria:

* Adult resident of the City of Lynchburg, Virginia
* Under-resourced at trial entry as defined by meeting eligibility for welfare, food stamps/SNAP, Medicaid, Housing Choice Voucher program, or income at or below 200% of the Federal Poverty Threshold.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Rides completed | 1 year
  Total number of rides for test subject per week, averaged over previous 6 months, measured at intake, 6 months, and 1 year.
Cost of transportation | 1 year
  Total cost per mile of transportation, averaged over previous 6 months, measured at intake, 6 months, and 1 year.
Untreated disease(s) | 1 year
  Total number of attributed disease diagnoses that are not being treated, measured at intake, 6 months, and 1 year.
Cancer screening success | 1 year
  Number of eligible cancer screening exams not performed (lung, colon, breast), measured at intake, 6 months, and 1 year.

SECONDARY OUTCOMES:
Unmet transportation needs | 1 year
  Total number of rides per week that test subject is unable to complete, averaged over 6 previous 6 months, measured at intake, 6 months, and 1 year.
Unmet medical transportation needs | 1 year
  Total number of medical (including mental health) appointments missed due to transportation, averaged over previous 6 months, measured at intake, 6 months, and 1 year.
Prescribed medications | 1 year
  Total number of prescribed medications, measured at intake, 6 months, and 1 year.
Prescribed medications not utilized | 1 year
  Total number of prescribed medications that are not being utilized (all cause), averaged over previous 6 months, measured at intake, 6 months, and 1 year.
Weight | 1 year
  Weight in pounds, measured at intake, 6 months, and 1 year.
BMI | 1 year
  Body mass index, measured at intake, 6 months, and 1 year.
Blood Pressure | 1 year
  Blood Pressure (mmHg), measured at intake, 6 months, and 1 year.
Hgb A1c | 1 year
  Hemoglobin A1c, measured at intake, 6 months, and 1 year.
ADL | 1 year
  Activities of daily living (Barthel index), measured at intake, 6 months, and 1 year.
IADL | 1 year
  Instrumental activities of daily living (Lawton scale), measured at intake, 6 months, and 1 year.
Physical activity | 1 year
  Physical activity / exercise assessment (Modified Kaiser physical activity survey), measured at intake, 6 months, and 1 year.
Psychosocial assessment | 1 year
  Psychosocial assessment (PAT, Briggs Health), measured at intake, 6 months, and 1 year.
Cognitive function | 1 year
  Cognitive function test (CPCOG), measured at intake, 6 months, and 1 year.
Depression screening | 1 year
  Depression screening and/or assessment (MHA depression screening tool), measured at intake, 6 months, and 1 year.
Other mental health conditions | 1 year
  Other mental health conditions (MHA screening and assessment tools), measured at intake, 6 months, and 1 year.
Smoking assessment | 1 year
  Smoking / tobacco / nicotine use (No/Yes, with yes triggering LDCT assessment), measured at intake, 6 months, and 1 year.
Substance use | 1 year
  Substance use or abuse (CAGE), measured at intake, 6 months, and 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: John Salmon, MD, Study Director — Medical Director, Lighthouse Community Health Center
Locations (1):
- Lighthouse Community Health Center, Lynchburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data from all three datasets
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available July 2024 (2 years)
Access Criteria: Government entity; Healthcare system

REFERENCES:
- [Background] Bradley EH, Elkins BR, Herrin J, Elbel B. Health and social services expenditures: associations with health outcomes. BMJ Qual Saf. 2011 Oct;20(10):826-31. doi: 10.1136/bmjqs.2010.048363. Epub 2011 Mar 29. PMID 21447501
- [Background] Solberg LI. Theory vs Practice: Should Primary Care Practice Take on Social Determinants of Health Now? No. Ann Fam Med. 2016 Mar;14(2):102-3. doi: 10.1370/afm.1918. No abstract available. PMID 26951583
- [Background] Hood CM, Gennuso KP, Swain GR, Catlin BB. County Health Rankings: Relationships Between Determinant Factors and Health Outcomes. Am J Prev Med. 2016 Feb;50(2):129-35. doi: 10.1016/j.amepre.2015.08.024. Epub 2015 Oct 31. PMID 26526164